CLINICAL TRIAL: NCT06163274
Title: MATRIX-003: Trial to Assess Acceptability and Safety of Two Placebo Intravaginal Ring Designs
Brief Title: Trial to Assess Acceptability and Safety of Two Placebo Intravaginal Rings
Acronym: MATRIX-003
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to Stop Work order issued on1/24/2025 as result of United States President's Executive Order on Reevaluating and Realigning United States Foreign Aid
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Oak Crest Institute of Science (Other)
Responsible Party: Principal Investigator, Catherine Anne Chappell, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY23070172
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Safety; Acceptability
Keywords: Vagina; Placebo; Intravaginal Ring

STUDY DESIGN:
Intervention Model Description: Participants will randomized to sequence of using 2 placebo intravaginal rings; Ring A followed by Ring B or Ring B followed by Ring A
Who Masked: Outcomes Assessor
Masking Description: The participants, care providers, and investigators may be able to tell the difference in the hardness/flexibility of the two rings after handling them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence: Placebo Intravaginal Ring A followed by Placebo Intravaginal Ring B (Experimental): Placebo Intravaginal Ring A will be inserted and used for 28 days, Ring A will be removed and followed by no intravaginal ring use for 7-21 days. Then Placebo Intravaginal Ring B will be inserted and used for 28 days.
  Interventions: Device: Placebo Intravaginal Ring A; Device: Placebo Intravaginal Ring B
- Sequence: Placebo Intravaginal Ring B followed by Placebo Intravaginal Ring A (Experimental): Placebo Intravaginal Ring B will be inserted and used for 28 days, Ring B will be removed and followed by no intravaginal ring use for 7-21 days. Then Placebo Intravaginal Ring A will be inserted and used for 28 days.
  Interventions: Device: Placebo Intravaginal Ring A; Device: Placebo Intravaginal Ring B

INTERVENTIONS:
Device: Placebo Intravaginal Ring A — Placebo Intravaginal Ring A consists of a flexible lavender silicone scaffold, with an outer diameter of 55 mm and a durometer value of 40A (Shore A hardness scale). The ring holds two blank grey cassettes.
Device: Placebo Intravaginal Ring B — Placebo Intravaginal Ring B consists of a flexible lavender silicone scaffold, with an outer diameter of 55 mm and a durometer value of 50A (Shore A hardness scale). The ring holds two blank grey cassettes.

SUMMARY:
This research study is being conducted to find out how easy, comfortable, and safe intravaginal rings are for women to use. The two rings used in this study do not dispense any medications, are the same size, but differ in their flexibility and hardness. This study will enroll approximately 100 HIV-negative persons, aged18-45 years, and assigned female sex at birth from sites in the United States, South Africa, and Zimbabwe. Participants will be randomly assigned to use (self-insert) Ring A for 4 weeks and then Ring B for 4 weeks or Ring B first followed by Ring A. There will be a 1-3-week rest period between using the two different rings. The study involves answering questions, undergoing pelvic examinations, and collecting blood and vaginal fluid samples over a total of 7 in-person visits and 2 telephone calls over approximately 9-11 weeks. In addition, both participants and approximately 30 of their sexual partners will be asked to take part in in-depth interviews to further assess acceptability, attitudes, and experiences with ring use to gauge interest in the future use of intravaginal rings as a HIV prevention option.

DETAILED DESCRIPTION:
The goal of this randomized, clinical trial is to compare two placebo intravaginal rings in HIV seronegative persons, aged 18-45 years, assigned female sex at birth who are at low risk of acquiring HIV infection. Participants will be recruited from five sites, one in the US and four in sub-Saharan Africa. Approximately 100 participants will be randomized (1:1), stratified by site, to the sequence of using the two intravaginal rings (A followed by B or B followed by A). The two rings differ only by mechanical attributes, such as flexibility and hardness. Each ring will be self-inserted and left in place for 4-weeks. After 4 weeks, the first assigned ring will be removed by the participant at the clinic. Then there will be a 7-21-day period of no ring use. The participant will then return to the clinic and self-insert the second assigned ring and leave it in place for 4 weeks, after which the participant will return to the clinic for self-removal of the ring. Differences in safety, acceptability, social harms and benefits, and composition of the vaginal microbiome between the two rings will be assessed. In addition, both participants and approximately 30 of their sexual partners will be asked to take part in in-depth interviews to further assess acceptability, attitudes, and experiences with ring use to gauge interest in the future use of intravaginal rings as a HIV prevention option.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female sex at birth.
* Able and willing to provide written informed consent to be screened for and enrolled in MATRIX-003 in one of the study languages.
* Able and willing to provide adequate contact/locator information.
* Able and willing to comply with all protocol requirements, including:

  * Abstaining from other intravaginal products or practices for the duration of the study.
  * Abstaining from penetrative vaginal intercourse (i.e., oral-, digital-, penile-penetration) for the first 14 days of each product use period.
  * Refraining from participation in other research studies involving drugs, medical devices, vaginal products, or vaccines starting 2 weeks before the Screening Visit and for the duration of the study, or in observational or qualitative studies for the duration of the study, unless approved by the Protocol Safety Review Team.
  * Reliable access to a private phone for scheduled phone contacts.
* HIV-uninfected based on testing performed at Screening and Enrollment.
* Per participant report, must be either not currently sexually active or in a mutually monogamous relationship with only one partner who is not known to be HIV positive or to currently have a sexually transmitted infection.
* Negative urine pregnancy test at Screening and Enrollment.
* Participants over the age of 21 (inclusive) must have documentation of a Grade 0 Pap smear within the past 3 years prior to Enrollment, or a Grade 1 Pap smear at Screening with no treatment required.
* Protected from pregnancy starting at least 2 weeks before Screening and continuing for the duration of study participation by an effective contraceptive method; effective methods include:

  * Hormonal methods except vaginal rings
  * Copper intrauterine device
  * Sterilization of participant or (if applicable) sterilization of monogamous partner
  * Correct and consistent condom use at study entry, and agrees to use site-provided condoms during study (for US site only)

Inclusion Criteria for sexual partner in-depth interview subset:

* Identifies as a sexual partner of a MATRIX-003 participant.
* Identified by participant as a sexual partner during MATRIX-003 for whom the participant has given permission to contact.
* Able and willing to provide written informed consent in one of the study languages.
* Able and willing to complete the required study procedures.
* Must be 18 years old or above at the time of their study participation.

Exclusion Criteria:

* Per participant report at Screening and Enrollment, intends to do any of the following during the study participation period:

  * Become pregnant.
  * Breastfeed.
  * Relocate away from the study site.
  * Travel away from the study site for a time period that would interfere with product resupply and/or study participation.
* Positive HIV test at Screening or Enrollment.
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, or Treponema pallidum (Syphilis) at Screening and (per participant report) treated for potential sexually transmitted infection within past 12 months.
* Diagnosed with urinary tract infection, pelvic inflammatory disease, or reproductive tract infection requiring treatment at Enrollment.

Note: Otherwise eligible participants diagnosed during screening with a urinary tract infection, symptomatic yeast infection or symptomatic bacterial vaginosis infection are offered treatment. If treatment is completed and symptoms have resolved within 45 days of obtaining informed consent for screening, the participant may be enrolled.

* Clinically apparent Grade 2 or higher pelvic exam finding at Enrollment.

Note: Otherwise eligible participants with exclusionary pelvic exam findings at Screening may be enrolled/randomized if treatment is completed at least 7 days prior to enrollment and findings have improved to a non-exclusionary severity grading or resolved by the time of enrollment. Spotting/bleeding will be considered exclusionary only if greater than what would be expected from contraceptive use.

* Participant report and/or clinical evidence of any of the following:

  * Known adverse reaction to silicone (ever).
  * Use of diaphragm, NuvaRing, or spermicide for contraception starting 2 weeks prior to Screening through Enrollment.
  * Use of any of the following in the past 12 months: stimulants (cocaine [including crack], methamphetamine, or non-physician prescribed pharmaceutical-grade stimulants), or inhaled nitrates, or illicit injection drug use of any kind.
  * Prior use of post-exposure prophylaxis or oral pre-exposure prophylaxis (including Emtricitabine/tenofovir) in the past 4 weeks or any prior use of long-acting systemic pre-exposure prophylaxis (including cabotegravir or islatravir).
  * Antibiotic, steroid, or antifungal (oral or intravaginal) therapy within 14 days of Enrollment.
  * Hysterectomy.
  * Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing, Intrauterine device insertion or removal, colposcopy) within 21 days prior to Enrollment.
  * At Screening or Enrollment, as determined by the Investigator of Record/designee, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease.
* Has any of the following laboratory abnormalities at Screening:

  * Grade 2 or higher Aspartate aminotransferase, alanine transaminase, creatinine, or Hemoglobin.
* Has any other condition that, in the opinion of the Investigator of Record/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants Preferring to Use Placebo Intravaginal Ring A versus Ring B | Through study completion, approximately 11 weeks
  Number of participants that report a preference to use placebo intravaginal Ring A versus Ring B
Mean Satisfaction with Placebo Intravaginal Ring Use | Through study completion, approximately 11 weeks
  Satisfaction will be assessed using a 10-point Likert scale with 0 being the least satisfied and 10 being the most satisfied

SECONDARY OUTCOMES:
Number of Participants with Genitourinary Grade 2 or Higher Adverse Events | Through study completion, approximately 11 weeks
  Number of participants with genitourinary Grade 2 or higher adverse events deemed related to placebo intravaginal ring use

OTHER OUTCOMES:
Mean Change in Nugent Score | Through study completion, approximately 11 weeks
  Mean change in the Nugent score as determined from vaginal smears. Nugent scores range from 0 to 10; 0 indicates a Lactobacillus-dominant microbiome while a score of 10 indicates a microbiome dominated by bacterial vaginosis-associated bacteria. Mean change will be assessed from pre-insertion and after 28 days of placebo intravaginal ring use for both rings A and B

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Chappell, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States
- South Africa (3):
  - Wits Reproductive Health and HIV Institute, Hillbrow, Johannesburg
  - Centre for the AIDS Programme of Research in South Africa - Vululindlela, Pietermaritzburg, KwaZulu-Natal
  - The Aurum Institue - Tembisa #4, Tembisa
- Harare Health and Research Consortium, Chitungwiza, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palanee-Phillips T, Baum MM, Moss JA, Clark MR, Nuttall J, Romano JW. Drug-releasing vaginal rings for HIV/STI and pregnancy prevention: a review of recent advances and clinical applications. Expert Opin Drug Deliv. 2022 Jan;19(1):47-58. doi: 10.1080/17425247.2022.2020242. Epub 2022 Jan 7. PMID 34958283
- [Background] Ridgeway K, Montgomery ET, Smith K, Torjesen K, van der Straten A, Achilles SL, Griffin JB. Vaginal ring acceptability: A systematic review and meta-analysis of vaginal ring experiences from around the world. Contraception. 2022 Feb;106:16-33. doi: 10.1016/j.contraception.2021.10.001. Epub 2021 Oct 10. PMID 34644609
- [Background] Stoner MCD, Browne EN, Gundacker HM, Hawley I, Chen BA, Hoesley C, Scheckter R, Piper J, Singh D, Song M, Liu A, van der Straten A. Acceptability of an extended duration vaginal ring for HIV prevention and interest in a multi-purpose ring. PLoS One. 2022 Feb 22;17(2):e0263664. doi: 10.1371/journal.pone.0263664. eCollection 2022. PMID 35192655
- [Background] Minnis AM, Etima J, Musara P, Browne EN, Mutero P, Kemigisha D, Mgodi NM, Nakabiito C, Shapley-Quinn MK, Stoner MCD, Hartmann M, Macagna N, Piper J, van der Straten A. Couples' Preferences for "2 in 1" Multipurpose Prevention Technologies to Prevent Both HIV and Pregnancy: Results of a Discrete Choice Experiment in Uganda and Zimbabwe. AIDS Behav. 2022 Dec;26(12):3848-3861. doi: 10.1007/s10461-022-03713-6. PMID 35674885

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT06163274/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT06163274/ICF_001.pdf